CLINICAL TRIAL: NCT04659187
Title: "CORONA Germany" - Clinical Outcome and Risk in Hospitalized COVID-19 Patients - An Epidemiological Study From Germany
Brief Title: CORONA Germany- Clinical Outcome and Risk in Hospitalized COVID-19 Patients - An Epidemiological Study From Germany
Acronym: CORONA Germany
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asklepios proresearch (Industry)
Collaborators: Asklepios Kliniken GmbH & Co. KGaA (Unknown)
Responsible Party: Sponsor
Other Study IDs: #3871
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: COVID-19; Corona; Risk factor; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- All hospitalized COVID-19 patients: All consecutive hospitalized patients, tested positive for SARS-CoV-2 at 45 Asklepios hospitals in Germany
- Subgroup: Detailed cohort of 7 hospitals: Cohort of 7 hospitals with detailed data set
- Subgroup with cardiovascular events: Definition: Patients hospitalized to COVID-19, who developed a cardiovascular event, defined as (1) cardiopulmonary resuscitation in cardiac arrest, (2) cardiogenic shock, (3) acute coronary artery syndrome, including ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI), (4) acute myocarditis, (5) denovo cardiac arrhythmia, (6) arterial or venous thrombosis, (7) pulmonary artery embolism, (8) worsening of prior or new onset heart failure, (9) ischemic stroke
- Subgroup with oncological patients: Definition: Patients hospitalized to COVID-19 with prior or preexisting oncological disease
- Subgroup with critical ill COVID-19 patients: Definition: Patients hospitalized to COVID-19 with intensive care treatment

SUMMARY:
This is a multicenter, observational, prospective, epidemiological cohort study at 45 hospitals in Germany, all part of a German hospital network. All hospitalized patients tested positive for SARS-CoV-2 will be included.

DETAILED DESCRIPTION:
CORONA Germany is a multicenter, observational, prospective, epidemiological cohort study at 45 hospitals in Germany, all part of a German hospital network. From January 1st till November 17th, 2020, all hospitalized patients tested positive for SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) will be included. Demographical data and outcomes will be assessed in the entire study cohort. In a subgroup, consisting of 7 hospitals, further detailed data (e.g. baseline characteristics, laboratory values, medication, clinical events) will be assessed. Additionally, there will be subgroups of patients with cardiovascular events and prior or preexisting oncological diseases. There are two primary endpoints: 1. Combination of all-cause death and/or need for mechanical ventilation and/or allocation to intensive care unit (ICU). 2. Occurrence of a clinical manifest cardiovascular events. The aim of the study is the development of a prediction model for the primary endpoints, whereas the secondary endpoint is a comparison of mortality rates between the 1st (01/01/20-09/15/20) and 2nd (15/09/20) infection wave. All endpoints will be verified by an Endpoint Review Committee. A Steering Committee, consisting of representatives of the 45 hospitals, the trial statistician and members of the scientific department, takes responsibility of the study design and results.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients tested positive for SARS CoV-2 using a reliable test method (mostly polymerase chain reaction test)

Exclusion Criteria:

* Patients with negative SARS CoV-2 testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive hospitalized patients tested positive for SARS CoV-2 using a reliable test method (mostly polymerase chain reaction test)
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-03-26 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite of death and/or need for mechanical ventilation and/or admission to ICU | 9 months
  Composite of death and/or need for mechanical ventilation and/or admission to ICU in patients hospitalized to COVID 19
Occurrence of a clinical manifest cardiovascular event | 9 months
  Occurrence of a clinical manifest cardiovascular Event, defined as (1) cardiopulmonary resuscitation in cardiac arrest, (2) cardiogenic shock, (3) acute coronary artery syndrome, including ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI), (4) acute myocarditis, (5) denovo cardiac arrhythmia, (6) arterial or venous thrombosis, (7) pulmonary artery embolism, (8) worsening of prior or new onset heart failure, (9) ischemic stroke

SECONDARY OUTCOMES:
Overall mortality and mortality rate | 9 months
  Comparison of mortality rates between the 1st (01/01/20-09/15/20) and 2nd (15/09/20) infection wave
Risk stratification score to predict the primary endpoints | 9 months
  Risk stratification score to predict the primary endpoint in hospitalized COVID 19 patients in the subgroup of seven hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U Herborn, Prof. MD, Principal Investigator — Asklepios Kliniken GmbH & Co. KGaA
Locations (8):
- Germany (8):
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Wandsbek, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Asklepios Kliniken GmbH & Co. KGaA, Hamburg
  - Asklepios Klinik Nord, Hamburg
  - Asklepios Westklinikum Hamburg, Hamburg
  - Asklepios Klinik Altona, Hamburg

IPD SHARING:
Plan to Share IPD: No
Individual patient data will be collected anonymously. Sharing is not planned.

REFERENCES:
- [Derived] Dickow J, Gunawardene MA, Willems S, Feldhege J, Wohlmuth P, Bachmann M, Bergmann MW, Gesierich W, Nowak L, Pape UF, Schreiber R, Wirtz S, Twerenbold R, Sheikhzadeh S, Gessler N. Higher in-hospital mortality in SARS-CoV-2 omicron variant infection compared to influenza infection-Insights from the CORONA Germany study. PLoS One. 2023 Sep 27;18(9):e0292017. doi: 10.1371/journal.pone.0292017. eCollection 2023. PMID 37756299
- [Derived] Sievering AW, Wohlmuth P, Gessler N, Gunawardene MA, Herrlinger K, Bein B, Arnold D, Bergmann M, Nowak L, Gloeckner C, Koch I, Bachmann M, Herborn CU, Stang A. Comparison of machine learning methods with logistic regression analysis in creating predictive models for risk of critical in-hospital events in COVID-19 patients on hospital admission. BMC Med Inform Decis Mak. 2022 Nov 28;22(1):309. doi: 10.1186/s12911-022-02057-4. PMID 36437469
- [Derived] Gessler N, Gunawardene MA, Wohlmuth P, Arnold D, Behr J, Gloeckner C, Herrlinger K, Hoelting T, Pape UF, Schreiber R, Stang A, Wesseler C, Willems S, Arms C, Herborn CU. Clinical outcome, risk assessment, and seasonal variation in hospitalized COVID-19 patients-Results from the CORONA Germany study. PLoS One. 2021 Jun 17;16(6):e0252867. doi: 10.1371/journal.pone.0252867. eCollection 2021. PMID 34138888